CLINICAL TRIAL: NCT03402945
Title: A Cluster-randomized Factorial Crossover Trial, Comparing Antibiotic Mono-prophylaxis With Cefazolin vs. Dual-prophylaxis With Cefazolin Plus Vancomycin and Conventional Wound Dressing vs. Prevena Negative-pressure Wound Management
Brief Title: Prevention of Infections in Cardiac Surgery (PICS) Prevena Study
Acronym: PICS-Prevena
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PICS-PREVENA V1_20171106
Record Dates: First submitted 2018-01-08; First posted 2018-01-18 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Surgical Site Infections
Keywords: negative pressure wound management system; open-heart surgery; antibiotic prophylaxis; surgical site infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Cefazolin; Vancomycin

STUDY DESIGN:
Intervention Model Description: 1) cefazolin prophylaxis plus Prevena*(*diabetic and/or obese patients (BMI >30kg/m2)) 2) cefazolin and vancomycin prophylaxis plus Prevena*(*diabetic and/or obese patients (BMI >30kg/m2)), 3) cefazolin prophylaxis plus standard wound dressing, 4) cefazolin and vancomycin prophylaxis plus standard wound dressing.
Who Masked: Outcomes Assessor
Masking Description: Blinded adjudication of the s-SSIs will be performed by a committee consisting of three members.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1 (Active Comparator): cefazolin prophylaxis plus Prevena negative-pressure wound management system . Cefazolin 2g (or 3g if greater than 120kg body weight) will be given within an hour of surgery, followed by one intra-operative dose of cefazolin at 4 hours after the first dose or upon wound closure (whatever comes first), and finally two post-operative doses q8h.
  Prevena will be applied to all diabetic and/or obese patients (BMI >30kg/m2) at the end of surgery on the sternal as well as the vein harvest site (if open saphenous vein harvest) in the OR and left in place for 7 day
  Interventions: Device: Prevena; Drug: Cefazolin
- Arm 2 (Active Comparator): cefazolin and vancomycin prophylaxis plus Prevena negative-pressure wound management system. Cefazolin 2g (or 3g if greater than 120kg body weight) within an hour of surgery, followed by one intra-operative dose of cefazolin at 4 hrs after the first dose or upon wound closure (whatever comes first), and finally two post-operative doses q8h. Vancomycin at roughly 15mg/kg body weight intravenously, i.e. 1g, or 1.5g if greater than 85kg body weight. No intra-operative dose of vancomycin will be given, and a single second dose will be given 12 hours after the first dose.
  Prevena will be applied to all diabetic and/or obese patients (BMI >30kg/m2) at the end of surgery on the sternal as well as the vein harvest site (if open saphenous vein harvest) in the OR and left in place for 7 days.
  Interventions: Device: Prevena; Drug: Cefazolin; Drug: Vancomycin
- Arm 3 (Active Comparator): cefazolin prophylaxis plus standard wound dressing. Cefazolin 2g (or 3g if greater than 120kg body weight) within an hour of surgery, followed by one intra-operative dose of cefazolin at 4 hours after the first dose or upon wound closure (whatever comes first), and finally two post-operative doses q8h.
  Standard wound dressing: non-negative wound dressing as standard of care at the study site.
  Interventions: Drug: Cefazolin; Other: standard wound dressing
- Arm 4 (Active Comparator): cefazolin and vancomycin prophylaxis plus standard wound dressing. Cefazolin 2g (or 3g if greater than 120kg body weight) within an hour of surgery, followed by one intra-operative dose of cefazolin at 4 hours after the first dose or upon wound closure (whatever comes first), and finally two post-operative doses q8h. Vancomycin at roughly 15mg/kg body weight intravenously, i.e. 1g, or 1.5g if greater than 85kg body weight. No intra-operative dose of vancomycin will be given, and a single second dose will be given 12 hours after the first dose.
  Standard wound dressing: non-negative wound dressing as standard of care at the study site.
  Interventions: Drug: Cefazolin; Drug: Vancomycin; Other: standard wound dressing

INTERVENTIONS:
Device: Prevena — Negative-Pressure Wound Management System
  Arms: Arm 1; Arm 2
Drug: Cefazolin — antibiotic
Drug: Vancomycin — antibiotic
  Other Names: Vancocin
  Arms: Arm 2; Arm 4
Other: standard wound dressing — Any non-negative pressure wound dressing that is routinely used at study sites will be considered standard of care in the control arms.
  Arms: Arm 3; Arm 4

SUMMARY:
This vanguard study will be conducted at two study sites in Canada. It is a cluster randomized trial to test a combination of two antibiotics for antibiotic prophylaxis as compared to routine prophylaxis with one single antibiotic, and to test a negative-pressure wound management system (Prevena) versus standard wound dressing to reduce chest wound infections.

DETAILED DESCRIPTION:
Despite the routine use of antibiotics before and after cardiac surgery, infections of the chest wound remain a common life threatening complication of heart surgery that is preventable. Antibiotic prophylaxis is well accepted to be the cornerstone of prevention for these infections. The best choice of antibiotic prophylaxis in patients undergoing open heart surgery is, however, unclear. A large number of relevant pathogens are not covered by the primarily recommended antibiotic for prophylaxis, and there is a large variability in the antibiotics physicians use in practice and a lack of evidence supporting these choices. Appropriate management of the wound is probably also highly relevant in terms of infection prevention; however, there is a lack of strong evidence guiding the choice of wound management strategies as a means to reduce surgical site infection. The proposed study will test whether dual antibiotic prophylaxis is superior to single-agent prophylaxis with cefazolin, and shed light on whether or not modern negative-pressure wound management technology lower the risk of sternal surgical site infections.

ELIGIBILITY:
Inclusion Criteria:

- ≥18 years of age undergoing open-heart surgery (sternotomy, including minimally-invasive sternotomies)

Exclusion Criteria:

* On systemic antibiotics or with an active bacterial infection at the time of surgery
* Patients previously enrolled in this trial
* Patients known to be colonized with Methicillin-resistant S. aureus (MRSA)(unethical not to administer glycopeptides), beta-lactam or vancomycin allergy precluding the use of cefazolin or vancomycin, respectively, or to silver precluding the use of Prevena
* Participation in other studies that may interfere with this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4107 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Adherence to the wound management system | Prevena or standard wound dressing applied after surgery as per protocol, assessed up to 90 days after surgery
  goal is >90%
Adherence to the antibiotic regimen | Cefazolin: within an hour of surgery; one intra-operative dose at 4 hours after the first dose or upon wound closure (whatever comes first); two post-operative doses q8h. Vancomycin: initially intravenously; second dose 12 hrs after the first dose.
  goal is >90%
Loss of follow-up | up to 90 days after surgery
  goal is <10%

SECONDARY OUTCOMES:
Deep incisional and organ/space sternal-surgical site infection (s-SSI) | up to 90 days after surgery
  using standardized CDC/NHSN (Centre for Disease Control and Prevention/National Healthcare Safety Network) definitions
Wound dehiscence | up to 90 days after surgery
  using standardized CDC/NHSN (Centre for Disease Control and Prevention/National Healthcare Safety Network) definitions
C. difficile infection | up to 90 days after surgery
  laboratory confirmed
Mortality in patients with an active infection | up to 90 days after surgery
  using standardized CDC/NHSN (Centre for Disease Control and Prevention/National Healthcare Safety Network) definitions
ICU (Intensive Care Unit) and hospital stay | Length of ICU - from date of surgery to initial ICU discharge date, assessed up to 90 days after surgery. Hospital Stay - date of surgery to date of hospital discharge, assessed up to 90 days after surgery.
  length
Pain on day 7 | Pain at Day 7 (+/- 1 day)
  Visual analog scale (VAS)
Acute kidney injury | within 7 days of surgery
  Based on serum creatinine, following Acute Kidney Injury Network definition

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Mertz, MD,MSc, Principal Investigator — Juravinski Hospital and Cancer Centre
Locations (2):
- Canada (2):
  - Hamilton General Hospital, Hamilton, Ontario
  - London Health Sciences Centre & Lawson Health Research Institute, London, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Connolly SJ, Philippon F, Longtin Y, Casanova A, Birnie DH, Exner DV, Dorian P, Prakash R, Alings M, Krahn AD. Randomized cluster crossover trials for reliable, efficient, comparative effectiveness testing: design of the Prevention of Arrhythmia Device Infection Trial (PADIT). Can J Cardiol. 2013 Jun;29(6):652-8. doi: 10.1016/j.cjca.2013.01.020. PMID 23702356
- [Background] Mertz D, Whitlock R, Kokoszka AY, Smith SW, Carignan A, Rehan M, Jaffer IH, Alsagheir A, Loeb M. Routine Surveillance Versus Independent Assessment by an Outcome Adjudication Committee in Assessing Patients for Sternal Surgical Site Infections After Cardiac Surgery. Infect Control Hosp Epidemiol. 2016 May;37(5):600-2. doi: 10.1017/ice.2015.347. Epub 2016 Jan 19. PMID 26782707
- [Background] Filsoufi F, Castillo JG, Rahmanian PB, Broumand SR, Silvay G, Carpentier A, Adams DH. Epidemiology of deep sternal wound infection in cardiac surgery. J Cardiothorac Vasc Anesth. 2009 Aug;23(4):488-94. doi: 10.1053/j.jvca.2009.02.007. Epub 2009 Apr 19. PMID 19376733
- [Background] Edwards FH, Engelman RM, Houck P, Shahian DM, Bridges CR; Society of Thoracic Surgeons. The Society of Thoracic Surgeons Practice Guideline Series: Antibiotic Prophylaxis in Cardiac Surgery, Part I: Duration. Ann Thorac Surg. 2006 Jan;81(1):397-404. doi: 10.1016/j.athoracsur.2005.06.034. No abstract available. PMID 16368422
- [Background] Lador A, Nasir H, Mansur N, Sharoni E, Biderman P, Leibovici L, Paul M. Antibiotic prophylaxis in cardiac surgery: systematic review and meta-analysis. J Antimicrob Chemother. 2012 Mar;67(3):541-50. doi: 10.1093/jac/dkr470. Epub 2011 Nov 13. PMID 22083832
- [Background] Mertz D, Johnstone J, Loeb M. Does duration of perioperative antibiotic prophylaxis matter in cardiac surgery? A systematic review and meta-analysis. Ann Surg. 2011 Jul;254(1):48-54. doi: 10.1097/SLA.0b013e318214b7e4. PMID 21412147